CLINICAL TRIAL: NCT00835055
Title: Expression of Molecular Markers Before and After Neo-adjuvant Chemoradiotherapy in Rectal Cancer
Status: Withdrawn | Type: Observational
Why Stopped: never started several reasons
Sponsor: St. Claraspital AG (Other)
Responsible Party: Principal Investigator, Dr. Beatrice Kern, Dr.med, St. Claraspital AG
Other Study IDs: 43/05
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Rectal Cancer
Keywords: rectal cancer with neoadjuvant treatment; standardized clinical tests; tumor markers on tumor tissue
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine whether markers on tumor tissue may be an indicator for good response to neoadjuvant chemoradiotherapy in patients with rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced rectal cancer uT3 or uT4
* no distant metastasis
* neoadjuvant radiochemotherapy required

Exclusion Criteria:

* rejection of radiochemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: group is selected from a single institution ( community hospital)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Claraspital, Chirurgische Klinik, Basel, Switzerland